CLINICAL TRIAL: NCT01821300
Title: Cardiometabolic Risk and Obesity in Adolescents With Down Syndrome
Brief Title: Down Syndrome Metabolic Health Study
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 12-009233; 1R01HD071981-01A1 (NIH)
Record Dates: First submitted 2013-03-27; First posted 2013-04-01 (Estimated); Results first posted 2019-01-09 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Down Syndrome; Trisomy 21
Keywords: Down syndrome; Philadelphia; The Children's Hospital of Philadelphia; Body composition; Obesity; Cardiovascular
MeSH Terms: conditions — Down Syndrome; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood serum will be retained.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Down syndrome: No intervention occurred as this was a cross sectional observational study.
- Control: No intervention occurred as this was a cross sectional observational study.

SUMMARY:
The purpose of this research study is to determine which measures best capture cardiovascular disease (CVD) risk and type 2 diabetes (T2DM) risk in children and adolescents with Down syndrome (DS).

We hypothesize that DS is associated with worse cardiometabolic risk factors for a given body mass index compared to controls. This difference arises at least in part, from increased fat tissue.

DETAILED DESCRIPTION:
DS affects 1 per 800 births and is one of the most common causes of developmental disability in the US. Life expectancy for Down syndrome has increased significantly: estimated median survival in the US in 1997 was 49 years. DS is associated with an increased risk for obesity, with an estimated prevalence of 47-48% in adults and 30-50% in children with DS. Adolescents with DS are more likely to have increased adiposity compared to unaffected peers and may be at increased risk for obesity-related co-morbidities, such as type 2 diabetes and cardiovascular disease. How one defines obesity in DS is not clear. Individuals with DS have short stature and possibly increased adiposity, and the body mass index (BMI) used to define obesity for otherwise healthy populations may not accurately depict body fatness or capture cardiometabolic risk in DS.

Congenital heart disease (CHD) affects approximately 50% of individuals with DS; the National Institutes of Health Heart Lung and Blood Institute (NHLBI) Working Group on Obesity and Other Cardiovascular Risk Factors in Congenital Heart Disease highlighted the high prevalence of obesity in the setting of CHD, and called for studies to identify obesity measures that are more sensitive than BMI as well as studies of CVD risk prevention. Unfortunately, clinicians caring for obese adolescents with DS with or without CHD have little scientific evidence upon which to base guidance regarding cardiometabolic risk (CMR): data regarding CVD risk and prevalence of pre-diabetes and T2DM in obese adolescents with DS are lacking.

The measure of body fatness which best predicts CMR in DS is not known. We plan to compare BMI and other measures of body fatness in healthy controls and adolescents with DS to determine which measures best capture CVD and/or T2DM risk. These data will equip medical providers with the tools to better assess risk, initiate prevention measures, and guide screening in adolescents with DS.

ELIGIBILITY:
Inclusion Criteria:

* Both groups: Ages 10 - 20
* Both groups: Parental/guardian permission (informed consent) and if appropriate, child assent.
* Down syndrome group only: diagnosis of Down syndrome

Exclusion Criteria (both groups):

* Major organ system illness (such as leukemia), except for type 2 Diabetes
* Cyanotic congenital heart disease and/or pulmonary hypertension
* Medically unstable congenital heart disease
* Pregnancy
* Genetic syndrome known to affect glucose tolerance
* Familial hypercholesterolemia
* Currently treated with medications known to affect insulin sensitivity (other than diabetes agents in participants with type 2 diabetes)

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Participants will be recruited from primary care and speciality clinics, Trisomy 21 events, T21 interest groups, and referrals.
Sampling Method: Non-Probability Sample
Enrollment: 257 (Actual)
Dates: Start 2013-02; Primary Completion 2017-08-25 (Actual); Study Completion 2017-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Kelly, MD, MSCE, Principal Investigator — Children's Hospital of Philadelphia
Locations (2):
- United States (2):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Magge SN, Zemel BS, Pipan ME, Gidding SS, Kelly A. Cardiometabolic Risk and Body Composition in Youth With Down Syndrome. Pediatrics. 2019 Aug;144(2):e20190137. doi: 10.1542/peds.2019-0137. Epub 2019 Jul 17. PMID 31315916
- [Derived] Kelly A, Magge SN, Walega R, Cochrane C, Pipan ME, Zemel BS, Cohen MS, Gidding SS, Townsend R. Cross-Sectional Study of Arterial Stiffness in Adolescents with Down Syndrome. J Pediatr. 2019 Sep;212:79-86.e1. doi: 10.1016/j.jpeds.2019.04.059. Epub 2019 Jun 11. PMID 31201031
- [Derived] Kelly A, Gidding SS, Walega R, Cochrane C, Clauss S, Townsend RR, Xanthopoulos M, Pipan ME, Zemel BS, Magge SN, Cohen MS. Relationships of Body Composition to Cardiac Structure and Function in Adolescents With Down Syndrome are Different than in Adolescents Without Down Syndrome. Pediatr Cardiol. 2019 Feb;40(2):421-430. doi: 10.1007/s00246-018-2014-5. Epub 2018 Nov 1. PMID 30386863
- [Derived] Xanthopoulos MS, Walega R, Xiao R, Prasad D, Pipan MM, Zemel BS, Berkowitz RI, Magge SN, Kelly A. Caregiver-Reported Quality of Life in Youth with Down Syndrome. J Pediatr. 2017 Oct;189:98-104.e1. doi: 10.1016/j.jpeds.2017.06.073. Epub 2017 Jul 24. PMID 28751125

RESULTS

PARTICIPANT FLOW:
Groups:
- Down Syndrome: 154 participants ages 10-20 years old.
  No intervention occurred as this is a cross-sectional observational study.
- Control: 103 age-, sex-, race-, ethnicity-, and BMI percentile-matched control subjects.
  No intervention occurred as this is a cross-sectional observational study.
Period: Overall Study
Arm/Group | Down Syndrome | Control
Started | 154 | 103
Completed | 154 | 103
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants from the Down syndrome and control groups were matched on BMI percentile, age, race, ethnicity, and sex.
Groups:
- Down Syndrome: Our goal is to enroll 155 subjects with Down syndrome, and to compare their data to our control group.
- Control: Our goal is to enroll 105 typically developing controls, who are matched to the Down syndrome group by age, sex, race, ethnicity, and BMI-z score.
- Total: Total of all reporting groups
Arm/Group | Down Syndrome | Control | Total
Number analyzed (Participants) | 154 | 103 | 257
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.4 (0.3) | 14.7 (0.3) | 14.7 (0.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 61 | 148
  Male | 67 | 42 | 109
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 6 | 19
  Not Hispanic or Latino | 141 | 97 | 238
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 30 | 24 | 54
  White | 117 | 74 | 191
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 3 | 4 | 7
Region of Enrollment [Number; unit: participants]
  United States | 154 | 103 | 257
BMI Percentile [Mean (Standard Deviation); unit: percentile] — Height & weight were measured and entered into the online CDC BMI Calculator for children and teens to determine percentile.
  percentile | 81.4 (1.8) | 79.3 (2.5) | 80.5 (1.4)

OUTCOME MEASURES:

1. Primary Outcome: Non-HDL Cholesterol
Description: Non-HDL cholesterol measured via fasting blood draw
Time Frame: Study Visit 1
Population: Participants excluded from lipid analysis if they failed to complete blood draw or were diagnosed with Type 1 Diabetes: DS=7, Controls=0
Measure: Median (Inter-Quartile Range); unit: mg/dl
Groups:
- Down Syndrome: Down syndrome participants in observational study.
- Control: Control participants in observational study.
Arm/Group | Down Syndrome | Control
Number analyzed (Participants) | 147 | 103
mg/dl | 128 [104 to 153] | 107 [92 to 123]

2. Primary Outcome: Lipid Subparticles
Description: Lipoprotein subclass particle analysis run on samples from fasting blood drawn Study Visit 1.
Time Frame: Study Visit 1
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: nmol/L
Arm/Group | Down Syndrome | Control
Number analyzed (Participants) | 147 | 103
nmol/L
  Small HDL-P (nmol/L) | 9.8 [5.3 to 14] | 11.7 [8.9 to 14.9]
  Large VLDL-P (nmol/L) | 3.9 [2.3 to 5.7] | 2.4 [1.5 to 4.1]
  Small LDL-P (nmol/L) | 518 [401 to 639] | 420 [315 to 529]
  Total LDL-P (nmol/L) | 977 [806 to 1193] | 850 [693 to 997]

3. Primary Outcome: Lipid Subparticles (Size)
Description: Lipoprotein subclass particle analysis run on samples from fasting blood drawn Study Visit 1.
Time Frame: Study Visit 1
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: nm
Arm/Group | Down Syndrome | Control
Number analyzed (Participants) | 147 | 103
nm
  HDL-P size (nm) | 9.6 [9.2 to 9.9] | 9.6 [9.1 to 9.9]
  VLDL-P size (nm) | 49.2 [45.8 to 53.6] | 47.1 [44.2 to 50.7]
  LDL-P size (nm) | 20.7 [20.3 to 21.2] | 20.7 [20.2 to 21.1]

4. Primary Outcome: Insulin Resistance
Description: Insulin Resistance (HOMA-IR) was calculated as [fasting insulin (uIU/mL) x fasting glycemia (mmol/L)]/22.5
Time Frame: Study Visit 1
Population: Participants excluded from insulin resistance analysis if they failed to complete blood draw or were diagnosed with Type 1 Diabetes: DS=147, Controls=103.
Measure: Median (Inter-Quartile Range); unit: HOMA-IR
Arm/Group | Down Syndrome | Control
Number analyzed (Participants) | 147 | 103
HOMA-IR | 1.8 [1.0 to 2.7] | 1.95 [0.92 to 3.4]

5. Primary Outcome: Cardiometabolic Risk Biomarker Proteins
Description: hs-CRP, PAI-1, and IL-6 run on samples from fasting blood drawn Study Visit 1.
Time Frame: Study Visit 1
Population: Participants excluded from analysis if they failed to complete blood draw or were diagnosed with Type 1 Diabetes: DS=7, Controls=0.
Measure: Median (Inter-Quartile Range); unit: ng/dL
Arm/Group | Down Syndrome | Control
Number analyzed (Participants) | 147 | 103
ng/dL
  IL-6 | 2.3 [1.4 to 3.5] | 1.5 [1.4 to 2.9]
  PAI-1 | 0.0204 [0.0132 to 0.0327] | 0.0254 [0.0147 to 0.0385]
  hs-CRP | 2.5 [0.64 to 6.9] | 1.0 [0.32 to 4.5]

6. Primary Outcome: Abnormal Glucose Tolerance
Description: Impaired fasting glucose (IFG) was defined as fasting glucose ≥ 100 mg/dl. Impaired glucose tolerance (IGT) was defined as 2-hour glucose 140-199 mg/dl measured as part of an oral glucose tolerance test.
Time Frame: Study Visit 1
Population: Participants completed an oral glucose tolerance test if they were in the overweight or obese categories: DS n=96, Control n=64.
Measure: Count of Participants; unit: Participants
Groups:
- Down Syndrome (Overweight & Obese Only): Down syndrome participants in observational study.
- Control (Overweight Obese Only): Control participants in observational study.
Arm/Group | Down Syndrome (Overweight & Obese Only) | Control (Overweight Obese Only)
Number analyzed (Participants) | 96 | 64
Participants
  Impaired Fasting Glucose | 12 | 3
  Abnormal Glucose Tolerance | 10 | 3

7. Primary Outcome: Visceral Fat
Description: Adiposity measured by Dual-energy X-ray absorptiometry
Time Frame: Study Visit 1
Measure: Median (Inter-Quartile Range); unit: cm^2
Arm/Group | Down Syndrome | Control
Number analyzed (Participants) | 154 | 103
cm^2 | 54.5 [39.9 to 81.9] | 55.9 [40.6 to 95.3]

8. Primary Outcome: Body Mass Measures
Description: Adiposity measured by Dual-energy X-ray absorptiometry
Time Frame: Study Visit 1
Measure: Median (Inter-Quartile Range); unit: g
Arm/Group | Down Syndrome | Control
Number analyzed (Participants) | 154 | 103
g
  Whole Body Fat Mass | 18607.5 [12034.8 to 27557.7] | 22372.1 [16143 to 39723.8]
  Whole Body Lean Mass | 34927.16 [27527.39 to 42383.86] | 44108.3 [32439.9 to 52181.3]

9. Primary Outcome: Left Ventricular Mass
Description: Cardiac end organ injury assessed by echocardiography. Left Ventricular Mass (LVM) was measured by area/length method using the apical four-chamber and parasternal short-axis views. LVM was calculated as LV area × LV length × 1.05 × 5/6.
Time Frame: Study Visit 1
Population: LVM was available in 136 adolescents with DS (60M/76F) and 101nonDS controls (41M/60F).
Measure: Median (Inter-Quartile Range); unit: g
Arm/Group | Down Syndrome | Control
Number analyzed (Participants) | 136 | 101
g | 68.3 [32.1 to 135] | 64 [53 to 77]

10. Primary Outcome: Pulse Wave Velocity
Description: Cardiac end organ injury assessed by Pulse Wave Velocity (PWV)
Time Frame: Study Visit 1
Population: PWV was available in 129 adolescents with DS and 97 controls
Measure: Median (Inter-Quartile Range); unit: m/s
Arm/Group | Down Syndrome | Control
Number analyzed (Participants) | 129 | 97
m/s | 5 [4.5 to 5.6] | 4.9 [4.5 to 5.5]

11. Secondary Outcome: Health Related Quality of Life - PedsQL
Description: Caregiver-perception of his/her child's health-related QOL was assessed with the use of the parent-proxy report of the Pediatric Quality of Life Inventory (PedsQL) Version 4.0. Sub-scale scores are converted to a 0-100 scale so that greater scores indicate better QOL. Scale scores are computed as the sum of the items divided by the number of items answered (this accounts for missing data). If more than 50% of the items in the scale are missing, the scale score is not computed. The Physical Health Summary Score (8 items) is the same as the Physical Functioning Scale. To create the Psychosocial Health Summary Score (15 items), the mean is computed as the sum of the items divided by the number of items answered in the Emotional, Social, and School Functioning Scales.
Time Frame: Study Visit 1
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Down Syndrome, Obese; Control, Obese: For the Psychosocial risk factors secondary analysis Down Syndrome and Control Groups were further divided into Obese and Not Obese sub groups for analysis.
- Down Syndrome, Not Obese: Our goal is to enroll 155 subjects with Down syndrome, and to compare their data to our control group.
  For the Psychosocial risk factors secondary analysis Down Syndrome and Control Groups were further divided into Obese and Not Obese sub groups for analysis.
- Control, Not Obese: Our goal is to enroll 105 typically developing controls, who are matched to the Down syndrome group by age, sex, race, ethnicity, and BMI-z score.
  For the Psychosocial risk factors secondary analysis Down Syndrome and Control Groups were further divided into Obese and Not Obese sub groups for analysis.
Arm/Group | Down Syndrome, Obese | Down Syndrome, Not Obese | Control, Obese | Control, Not Obese
Number analyzed (Participants) | 63 | 87 | 24 | 34
score on a scale
  Physical Functioning (PedsQL) | 68.3 (18.5) | 73.2 (21.4) | 78.9 (18.8) | 89.7 (19.7)
  Emotional (PedsQL) | 73.3 (76.0) | 76.0 (14.9) | 75.6 (19.5) | 77.2 (25.1)
  Social (PedsQL) | 60.7 (20.9) | 63.3 (19.2) | 80.4 (16.4) | 85.0 (22.3)
  School (PedsQL) | 65.1 (18.2) | 64.0 (17.2) | 75.6 (18.5) | 80.0 (24.0)
  Psychosocial (PedsQL) | 65.1 (14.3) | 67.8 (13.8) | 77.2 (15.4) | 80.7 (22.4)
  Total Score (PedsQL) | 66.2 (13.2) | 69.6 (14.2) | 77.8 (14.0) | 83.9 (21.0)

12. Secondary Outcome: Health Related Quality of Life - IWQOL
Description: Parent perception of the effects of weight on his/her child's QOL was assessed with a caregiver-proxy version of the Impact of Weight on Quality of Life - Kids (IWQOL-Kids) questionnaire. The IWQOL-Kids is a validated, 27-item, self-report measure of weight-related QOL for youth ages 11-19 years. It yields 4 subscales (Physical Comfort, Body Esteem, Social Life, and Family Relations) and a Total score, which have strong psychometric properties, discriminate among weight status groups, and are responsive to weight change. Scaled scores are standardized and range from 0 to 100, with greater scores representing better weight-related QOL.
Time Frame: Study Visit 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Down Syndrome, Obese | Down Syndrome, Not Obese | Control, Obese | Control, Not Obese
Number analyzed (Participants) | 63 | 87 | 24 | 34
score on a scale
  Physical Comfort (IWQOL-Kids) | 83.3 (18.6) | 97.1 (7.5) | 86.0 (16.6) | 98.2 (7.9)
  Body Esteem (IWQOL-Kids) | 91.4 (11.1) | 98.0 (5.4) | 73.9 (25.7) | 93.9 (12.8)
  Social Life (IWQOL-Kids) | 89.7 (17.6) | 98.4 (5.9) | 80.7 (21.0) | 95.0 (14.0)
  Family Relationships (IWQOL-Kids) | 93.8 (13.5) | 98.6 (5.3) | 93.2 (11.2) | 97.5 (8.9)
  Total (IWQOL-Kids) | 89.8 (11.7) | 98.0 (5.1) | 82.4 (16.7) | 95.9 (10.5)

ADVERSE EVENTS:
Time Frame: Adverse Events are monitored throughout participants' roughly 6 hour study visit, and for the 2 weeks following study visit while participants are wearing accelerator armbands and completing dietary recalls at home.
Arm/Group | Down Syndrome | Control
All-Cause Mortality (participants affected / at risk) | 0/154 | 0/103
Serious Adverse Events (participants affected / at risk) | 0/154 | 0/103
Other Adverse Events (participants affected / at risk) | 7/154 | 3/103
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Down Syndrome (N=154) | Control (N=103)
Skin irritation (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (2) — Skin irritation due to physical activity armband wear. If irritation occurred armband wear was discontinued.
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) — Vomiting in reaction to glucola ingestion associated with oral glucose tolerance test.
Fainting (General disorders) | 0 (0) | 1 (1) — Fainting in reaction to blood draw.
Hypoglycemia (Endocrine disorders) | 1 (1) | 0 (0) — Hypoglycemia occurring during oral glucose tolerance test. Test prematurely stopped so that participant could ingest food.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-21): https://cdn.clinicaltrials.gov/large-docs/00/NCT01821300/Prot_SAP_000.pdf